CLINICAL TRIAL: NCT00886197
Title: Diagnostic Efficacy of Narrow Band Imaging (NBI) in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Diagnostic Efficacy of Narrow Band Imaging in Patients With Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yi-Chia Lee, National Taiwan University Hospital
Other Study IDs: 200707042R
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: reflux; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GERD: 1. Symptomatic reflux subjects who receive esophagogastroscopy, aged from 20 to 70 years old.
  2. Patients with typical reflux symptoms (heartburn and/or acid regurgitation) at least 3 times per week in recent 4 months.

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common disorder in Asia that includes erosive and non-erosive counterparts. The evaluation of intra-esophageal damage is of paramount importance because patients with erosive and those with non-erosive GERD have distinct manifestations and prognoses. Although proton-pump inhibitor (PPI) is the treatment of choice for erosive patients with excellent therapeutic response, the majority of reflux patients can be classified with non-erosive reflux disease (NERD).Narrow-band imaging (NBI) is a novel, noninvasive optical technique that adjusts reflected light to improve the contrast of capillary patterns compared with conventional illumination. Based on the standard procedure of sequential conventional white-light, NBI, and magnified NBI, the investigators have validated the reliability of the diagnostic testing. The investigators will also enroll NERD patients to test their therapeutic response to rabeprazole. The investigators can find out the best strategy to identify the PPI responder.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a common disorder in Asia that includes erosive and non-erosive counterparts. The evaluation of intra-esophageal damage is of paramount importance because patients with erosive and those with non-erosive GERD have distinct manifestations and prognoses. Although proton-pump inhibitor (PPI) is the treatment of choice for erosive patients with excellent therapeutic response, the majority of reflux patients can be classified with non-erosive reflux disease (NERD).1 Not all of them demonstrate a favorable response to PPI treatment because the pathogenesis of NERD is in part associated with psychosomatic pathways.2 Their therapeutic response to PPI is unpredictable. Therefore, how to improve the diagnosis of reflux-induced mucosal damage under endoscopy is a worthwhile endeavor.

Minimal change esophagitis is commonly accepted as part of the spectrum of reflux esophagitis in Japan.3,4 This category is defined as "erythema without sharp demarcation, whitish turbidity, and/or invisibility of vessels due to these findings".3 Although the minimal change disease (MCD) can be recognized in a significant number of patients with reflux using endoscopy-first policy, the major drawback of this category from the Los Angeles system is due to a poor interobserver agreement (κ statistic = 0.2).

Narrow-band imaging (NBI) is a novel, noninvasive optical technique that adjusts reflected light to improve the contrast of capillary patterns compared with conventional illumination.5 This system is highly applicable in the detection of early-stage mucosal lesions, including oral cancer, Barrett's esophagus, gastric cancer, and colonic neoplasm.6-10 For the reflux patients we face on a daily basis, the NBI system has been proven to improve the intraobserver and interobserver reproducibilities in grading esophagitis with small erosive foci (improving overall κ value to 0.62 versus 0.45).11 Corresponding to the crowding of capillaries, inflamed mucosal breaks appear dark brown on NBI, which produces intense contrast against the normal squamous epithelium and the stomach mucosa. These properties may improve our ability to delineate the margins of small inflammatory foci. Based on this advantage, we plausibly hypothesize the use of this system may improve the description of MCD and enable the prediction of therapeutic response to PPI. Testing this hypothesis is the main goal of our study.

Aim of the Study To assess the clinical utility and therapeutic implications of NBI in evaluating reflux patients with minimal mucosal damage.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic reflux subjects who receive esophagogastroscopy, aged from 20 to 70 years old.
2. Patients with typical reflux symptoms (heartburn and/or acid regurgitation) at least 3 times per week in recent 4 months.

Exclusion Criteria:

1. Symptomatic reflux patients with apparent erosive esophagitis in conventional endoscopy.
2. Symptomatic reflux patients with a history of using PPI in recent 4 months.
3. Subjects with known allergy to PPI.
4. Peptic ulcer disease
5. Cancers of the esophagus, stomach, and duodenum
6. Esophageal varices.
7. Active upper gastrointestinal bleeding within 7 days prior to enrollment
8. Status after total or subtotal gastrectomy
9. Use of anticoagulants or antiplatelets within one week prior to enrollment
10. Subjects with bleeding tendency

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Symptomatic reflux subjects who receive esophagogastroscopy, aged from 20 to 70 years old.
  2. Patients with typical reflux symptoms (heartburn and/or acid regurgitation) at least 3 times per week in recent 4 months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Therapeutic response to proton-pump inhibitor (PPI) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chia Lee, MD,MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan